CLINICAL TRIAL: NCT06063395
Title: Study of the Size of the Operating Fields Depending on the Morphology of the Patients
Acronym: ABORD-3D
Status: Completed | Type: Observational
Sponsor: Geprovas (Network)
Responsible Party: Sponsor
Other Study IDs: 2023-A01613-42
Record Dates: First submitted 2023-09-18; First posted 2023-10-02 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Open Surgery on the Abdominal Aorta
Keywords: Abdominal aorta; Open surgery; Vascular surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient undergoing open surgery on the abdominal aorta by laparotomy
  Interventions: Procedure: open surgery on the abdominal aorta by laparotomy

INTERVENTIONS:
Procedure: open surgery on the abdominal aorta by laparotomy — Laparotomy aortic surgery for the management of an abdominal aortic aneurysm has several distinct stages which will not be altered by the performance of this study. The patient arrives in the operating room and is taken care of by the anesthetic team. The patient is then placed in the correct position for optimal surgical management and a skin cleansing procedure is carried out. A sterile drape is applied and the preoperative checklist in force in the establishment is completed. Initial dissection of the aneurysm and its proximal and distal control is left to the discretion of the principal surgeon. Once the aortic aneurysm has been controlled, the main surgeon places self-static retractors and then prepares to clamp the aorta. The surgeon initiates aortic clamping to create the aorto-biliac or bifemoral bypass. Once the bypass has been created, the operation is completed by closing the surgical approach and the skin incision. The bandage is then applied.

SUMMARY:
This is a prospective, single-centre, observational clinical study.

Patients who have not expressed their non-opposition, who are of age and who are undergoing open surgery on the abdominal aorta by laparotomy will be included.

The aim is to mathematically model the working volume for abdominal aortic surgery as a function of the preoperative CT scan, the length and orientation of the incision and the morphometric characteristics of the patient, and thus predict the surgical risk.

To meet this objective, the dimensions of the working volume of open abdominal aortic surgery will be measured using a camera to create an algorithm by associating them with the preoperative images and morphometric data of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patient undergoing open surgery on the abdominal aorta by laparotomy.
* Patient who has been informed of the terms of the study and who has not expressed non-opposition.

Exclusion Criteria:

* Emergency surgery
* Patient without preoperative CT scan

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient undergoing open surgery on the abdominal aorta by laparotomy.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Mathematically model the working volume for abdominal aortic surgery as a function of the preoperative CT scan, the length and orientation of the incision and the morphometric characteristics of the patient, and thus predict surgical risk. | During surgery
  To measure the dimensions of the working volume of an open abdominal aortic surgery using a camera to create an algorithm by associating them with the preoperative images and morphometric data of the patient.

SECONDARY OUTCOMES:
Find a correlation between work volume and BMI du patient. | During surgery
  Coefficient of determination R² which measures the quality of prediction of work volume as a function of patient BMI
Validate the algorithm for predicting the volume of work in abdominal aortic abdominal aortic surgery. | During surgery
  Difference in cubic centimetres between the volume of work and the predicted one
Evaluation of how the algorithm helps to deal with surgery | During surgery
  Evaluation questionnaire for surgeons
Correlate results with surgical complications | During the procedure until patient discharge
  Intra-hospital complications

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Chakfe, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France, France